CLINICAL TRIAL: NCT03998137
Title: A Prospective, Controlled, Multi-Center, Post-Approval Trial to Evaluate the Long-term Safety and Effectiveness of AUGMENT® Injectable Bone Graft Compared to Autologous Bone Graft as a Bone Regeneration Device in Foot and Ankle Fusions
Brief Title: Long-term Safety and Effectiveness of AUGMENT® Injectable Bone Graft Compared to Autologous Bone Graft
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BMTI-2018-01
Record Dates: First submitted 2019-06-19; First posted 2019-06-26 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Ankle and Hindfoot Arthrodesis
Keywords: Ankle Fusions; AUGMENT® Injectable Bone Graft; Autologous Bone Graft; arthritis; ankle pain; foot pain; hindfoot fracture; ankle fracture
MeSH Terms: conditions — Arthritis; Ankle Fractures | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples for antibody testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Autograft: Standard Rigid Fixation plus autograft
  Interventions: Procedure: Standard of Care
- AUGMENT® Injectable: Standard rigid fixation plus AUGMENT® Injectable Bone Graft
  Interventions: Device: AUGMENT® Injectable Bone Graft

INTERVENTIONS:
Device: AUGMENT® Injectable Bone Graft — AUGMENT® Injectable Bone Graft
  Groups: AUGMENT® Injectable
Procedure: Standard of Care — Autologous Bone Graft
  Groups: Autograft

SUMMARY:
The objective of this long-term study is to evaluate the long-term effectiveness and safety of AUGMENT® Injectable Bone Graft vs. autologous bone graft. The study involves evaluation of subjects originally treated under protocol BMTI-2009-01 or BMTI-2010-01 or treated with autograft under protocol BMTI-2006-01.

Subjects will be asked to consent and return to provide long-term follow-up data at or after 60 months (5 years) have elapsed since their original surgery as a subject in protocol BMTI-2009-01 or BMTI-2010-01.

STUDY HYPOTHESIS: The effectiveness and safety profile for AUGMENT® Injectable Bone Graft is maintained and remains comparable to that of autologous bone graft over long-term subject follow-up.

REGULATORY PHASE: Post-approval study

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing and able to provide informed consent and be available for the planned follow-up evaluations and radiologic tests; and
2. Must have been included in the Augment Injectable propensity score matching population from the Augment Injectable summary of safety and effectiveness data (SSED).

Exclusion Criteria:

1) Subjects that were excluded from the safety analysis in the BMTI-2009-01 or BMTI-2010-01 study. These subjects were consented, but never treated as part of the BMTI-2009-01 or BMTI-2010-01 protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects over the age of 18 years of age, who were randomized and treated as part of the population of the BMTI-2009-01 or BMTI-2010-01 protocol.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pain on weight bearing via Visual Analog Scale (VAS) | Visit 1 (Day 0)
  Subjects were asked to stand and report pain on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).

SECONDARY OUTCOMES:
Confirmation of bridging bone via computerized tomography (CT) | Visit 1 (Day 0)
  Overall Assessment of Osseous Bridging (% Bone Bridging; CT Scans)
  * Absent (0-24%)
  * Minimal (25-49%)
  * Moderate (50-74%)
  * Complete (75-100%)
AOFAS (American Orthopaedic Foot & Ankle Society) Hindfoot and Ankle Score | Visit 1 (Day 0)
  Subjects were asked to report pain, functionality and ability levels while the physician performed assessments based on alignment, abnormality, motion, and stability. The total score ranges from a low of zero to a high of 100, with subscales measuring pain (40 points), function (50 points), and alignment (10 points), with higher scores showing better outcomes.
Foot Function Index, FFI | Visit 1 (Day 0)
  The Foot Function Index (FFI) measures the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales all ranging from 0-100. To obtain a sub-scale score, the item scores for a sub-scale are totaled and then divided by the maximum total possible for all of the sub-scale items which the subject indicated were applicable. Any item marked as not applicable is excluded from the total possible. Sub-scales are an average of the completed ratings within that sub-scale. The total foot function score is an average of the three sub-scale scores and ranges from 0-100. Lower scores are indicative of better outcomes whereas higher scores indicate greater impairment.